CLINICAL TRIAL: NCT03803241
Title: Cd133+ Cell Infusion in Patients With Colorectal Liver Metastases That Are Going to be Submitted to a Major Liver Resection
Brief Title: Cd133+ Cell Infusion in Patients With Colorectal Liver Metastases.
Acronym: cellcol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Alejandra Garcia Botella, Principal investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-001402-18
Record Dates: First submitted 2016-11-18; First posted 2019-01-14 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVE + CD133 (Experimental): preop portal vein embolization + stem cells infusion
  Interventions: Drug: CD133+ infusion; Other: portal vein embolization
- PVE (Sham Comparator): only preop portal vein embolization
  Interventions: Other: portal vein embolization

INTERVENTIONS:
Drug: CD133+ infusion — Infusion of cells cd133+
  Arms: PVE + CD133
Other: portal vein embolization — portal vein embolization

SUMMARY:
Treatment of patients with metastatic colorectal carcinoma is surgical resection. Only 10-15% of the patients will be candidates for curative resection. After response to chemotherapy this figure rises 10-13% more. To perform the surgery it is necessary to have a sufficient remnant liver volume (RLV), which allows maintaining optimal liver function after resection. If the estimated RLV is insufficient preoperatively, portal venous embolization site (PVE) is performed for compensatory hypertrophy, thus increasing the number of resections 19%. Still, in 20% of these patients surgery can not be performed because RLV is not achieved or because the disease progresses while waiting for growth. Therefore, it is necessary to improve liver regeneration without promoting tumor growth. Studies on liver regeneration, have determined that cells (CD133 +) are involved in the liver hypertrophy that occurs after hepatectomy. CD133 + have been used to induce liver hypertrophy with encouraging results. This population of CD133 +, can be selected from peripheral blood after stimulation with Granulocyte colony-stimulating factor (G-CSF), being able to obtain a large number of them. The investigators propose to treat patients who do not meet criteria for surgery because of insufficient volume <40%, with CD133 + and portal embolization in order to carry out a surgical resection in a second place.

ELIGIBILITY:
Inclusion criteria:

1. Men and women between ≥ 18 years and ≤ 80. Women in fertile age should use contraceptive methods recommended by the Clinical Trial Facilitation Group (CTFG).
2. ECOG (Eastern Cooperative Oncology Group) quality of life scale ≤ 2.
3. Patients with hepatic metastases of colorectal carcinoma and insufficient hepatic remnant function to perform a major hepatectomy. This volume would be calculated by Positron emission tomography-Computed tomography (PET-CT) images or 64-channel multidetector CT.

   In patients who have received preoperative chemotherapy, the estimate residual liver volume to be included in the study will be <40%.

   Patients who have preserved liver function (Child ≤ B7 and International Normalized Ratio (INR) ≤ 2 in non-anticoagulated patients) and those who have not received chemotherapy, needs < 30% of residual volume to be included in the study.
4. Patients should have signed informed consent.

Exclusion criteria:

1. Pregnancy or lactation period.
2. Any condition that the investigators consider an unjustifiable risk in the patient.
3. Severe comorbidities: American Society of Anesthesiologists (ASA) ≥ 4.
4. Alterations in the hemogram and morphological alterations, evaluated by hematologist prior to administration of G-CSF.
5. Liver function: Child ≥ B7 and INR ≥ 2 in non-anticoagulated patients. In anticoagulated patients the values will have to be reverse, prior to surgery.
6. Patients who have not received research drugs in the last 30 days or in the period of 5 elimination half-life.
7. In patients on chemotherapy treatment, G-CSF can not be administered until 48 hours after the last administration of chemotherapy. Patients who have received Bevacizumab must wait 30 days since the last administration.
8. In addition, all those aspects that prevent the patient from being part of the study, understand the rules, follow the instructions given, or other aspects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Liver volume | once residual liver volume reach >40%, an average of 5 weeks.
  Liver volume estimated by computed tomography

SECONDARY OUTCOMES:
Liver volume | Post-surgery follow-up visits the first 30 days
  Liver volume estimated by computed tomography
Liver volume | Post-surgery follow-up visits the first 90 days
  Liver volume estimated by computed tomography
Liver volume | Post-surgery follow-up visits the first 180 days
  Liver volume estimated by computed tomography
Liver volume | Post-surgery follow-up visits the first 12 months
  Liver volume estimated by computed tomography
Liver volume | Post-surgery follow-up visits the first 18 months
  Liver volume estimated by computed tomography
Liver volume | Post-surgery follow-up visits the first 24 months
  Liver volume estimated by computed tomography

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Clinico San Carlos, Madrid
  - Alejandra Garcia Botella, Madrid

REFERENCES:
- [Derived] Garcia-Botella A, Saez-Carlin P, Mendez R, Martin MP, Ortega L, Mendez JV, Garcia-Paredes B, Diez-Valladares L, Torres AJ. CD133 + cell infusion in patients with colorectal liver metastases going to be submitted to a major liver resection (CELLCOL): A randomized open label clinical trial. Surg Oncol. 2020 Jun;33:224-230. doi: 10.1016/j.suronc.2019.10.005. Epub 2019 Oct 7. PMID 32561087